CLINICAL TRIAL: NCT04984135
Title: Drug-coated Balloon Angioplasty for De-novo or in-Stent Restenotic Coronary Lesions: an Optical Coherence Tomography Analysis
Brief Title: DCB Angioplasty for Coronary Lesions: an OCT Analysis
Status: Completed | Type: Observational
Sponsor: The First Affiliated Hospital of Dalian Medical University (Other)
Responsible Party: Sponsor
Other Study IDs: YJ-KY-FB-2021-09
Record Dates: First submitted 2021-07-25; First posted 2021-07-30 (Actual); Last update posted 2021-08-16 (Actual); Status verified 2021-08

CONDITIONS: Coronary Stenosis; Drug-coated Balloon
Keywords: Drug-coated balloon; Optical coherence tomography; De-novo coronary lesions; In-stent restenosis
MeSH Terms: conditions — Coronary Stenosis | interventions — Percutaneous Coronary Intervention

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Enrolled patients: Patients fulfilling the study criteria were included.
  Interventions: Procedure: Percutaneous coronary intervention

INTERVENTIONS:
Procedure: Percutaneous coronary intervention — All patients were treated with a loading dose of clopidogrel 300 or 600 mg before the procedure followed by maintenance clopidogrel 75 mg daily for 6 months. 100 U/ kg of unfractionated heparin was injected intravenously to maintain an activated clotting time ≥ 250 s during the procedure. For DCB treatment, the patient underwent predilation with an optimal-sized balloon (non-compliant balloon or cutting balloon) based on angiography (balloon-to-vessel ratio of 1.0), with the standard balloon shorter than the intended DCB size. The DCB was sized at 1:1 balloon-to-vessel ratio, delivered rapidly (median of 15 s) and inflated at nominal pressure for 60 s.

SUMMARY:
In this study, the investigators preformed OCT before and after DCB treatment, as well as at 6 months of follow-up, to assess the tissue characterization. The aim of this study was to investigate the relationship between quantitative and qualitative OCT findings, angiographic and clinical outcomes after PCB for coronary lesions.

DETAILED DESCRIPTION:
The paclitaxel drug-coated balloon (DCB) is an emerging device in percutaneous coronary intervention (PCI); it allows a rapid local release of an anti-restenotic drug without the use of a durable polymer or metal scaffold. The DCB has been proven to be effective with paclitaxel in preclinical trials and in clinical practice for the treatment of coronary lesions such as in-stent restenosis (ISR), de novo and bifurcation lesions. Optical coherence tomography (OCT) is an intravascular imaging modality that has higher resolution than intravascular ultrasound. Excellent contrast among lumen, vessel, and stent in OCT images allows accurate measurement of lumen and lesion. However, only a few studies have investigated the effect of DCB on the intimal lumen in the acute phase and during the follow-up using optical coherence tomography (OCT). In this study, the investigators preformed OCT before and after DCB treatment, as well as at 6 months of follow-up, to assess the tissue characterization.

Demographic, angiographic, and procedural data were collected. Participants were followed up with coronary angiography and OCT for at least 6-9 months, combined with OCT to analyze qualitative analysis of changes in plaque characterization, and late lumen loss. The participants were followed up for long-term clinical events (including cardiac death, target vessel myocardial infarction, and clinically driven target lesion revascularization).

ELIGIBILITY:
Inclusion Criteria:

* Coronary angiography shows that at least one coronary artery has a diameter stenosis >70% (left main stem diameter stenosis>50%)
* Stable or unstable angina
* Availability for follow-up for up to 12 months

Exclusion Criteria:

* Acute myocardial infarction within 48 hours
* Severe calcified lesions
* Unable to tolerate dual antiplatelet treatment (DAPT)
* Severe abnormal hematopoietic system, such as platelet count of < 100×109/L or > 700×109/L and white blood cell count of < 3×109/L
* Active bleeding or bleeding tendency
* Severe coexisting conditions, such as severe renal insufficiency (GFR < 60 ml/min•1.73m2), severe hepatic dysfunction [elevated ALT (glutamicpyruvic transaminase) or AST (glutamic-oxal acetic transaminase) level by more than three-fold of the normal limitation], acute or chronic heart failure (NYHA III-IV), acute infectious diseases, immune disorders, malignancy, etc.
* Life expectancy < 12 months
* Pregnancy or planning pregnancy
* Drug allergies or contraindications to aspirin, clopidogrel, ticagrelor, statins, contract, anticoagulant, stent, etc.
* Participation or planning to participate in another clinical trial during the same period
* Refusal to comply with the study protocol

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with de-novo or in-stent restenotic coronary lesions were treated with DCB
Sampling Method: Non-Probability Sample
Enrollment: 70 (Actual)
Dates: Start 2020-12-01 (Actual); Primary Completion 2021-07-01 (Actual); Study Completion 2021-07-20 (Actual)

PRIMARY OUTCOMES:
In-segment late lumen loss | 6 months
  Changes to lumen area assessed with the use of OCT

SECONDARY OUTCOMES:
Target lesion failure | 6 months
  The secondary endpoint was the incidence of target lesion failure (TLF), a composite of cardiac death, target vessel myocardial infarction, and clinically driven target lesion revascularization (TLR) at 6 months.

CONTACTS AND LOCATIONS:
Overall Officials: Lei Guo, MD, Principal Investigator — The First Affiliated Hospital of Dalian Medical University
Locations (1):
- The First Affiliated Hospital of Dalian Medical University, Dalian, Liaoning, China

REFERENCES:
- [Result] Tada T, Kadota K, Hosogi S, Miyake K, Ohya M, Amano H, Izawa Y, Kanazawa T, Kubo S, Ichinohe T, Hyoudou Y, Hayakawa Y, Sabbah MM, Otsuru S, Hasegawa D, Habara S, Tanaka H, Fuku Y, Katoh H, Goto T, Mitsudo K. Association between tissue characteristics assessed with optical coherence tomography and mid-term results after percutaneous coronary intervention for in-stent restenosis lesions: a comparison between balloon angioplasty, paclitaxel-coated balloon dilatation, and drug-eluting stent implantation. Eur Heart J Cardiovasc Imaging. 2015 Oct;16(10):1101-11. doi: 10.1093/ehjci/jev031. Epub 2015 Mar 9. PMID 25762559
- [Result] Miura K, Tada T, Habara S, Kuwayama A, Shimada T, Ohya M, Murai R, Amano H, Kubo S, Otsuru S, Tanaka H, Fuku Y, Goto T, Kadota K. Optical Coherence Tomography Predictors for Recurrent Restenosis After Paclitaxel-Coated Balloon Angioplasty for Drug-Eluting Stent Restenosis. Circ J. 2018 Oct 25;82(11):2820-2828. doi: 10.1253/circj.CJ-18-0464. Epub 2018 Aug 30. PMID 30158345
- [Result] Fukushima T, Ashikaga T, Yoshikawa S, Hatano Y, Ueshima D, Yamamoto T, Yasuhiro M, Isobe M. Effect of drug-coated balloon on stent restenosis, neointimal proliferation, and coronary dissection: an optical coherence tomography analysis. Coron Artery Dis. 2018 Jan;29(1):39-45. doi: 10.1097/MCA.0000000000000552. PMID 28902718
- [Result] de la Torre Hernandez JM, Garcia Camarero T, Lozano Ruiz-Poveda F, Urbano-Carrillo CA, Sanchez Perez I, Cano-Garcia M, Saez R, Andres Morist A, Molina E, Pinar E, Torres A, Lezcano EJ, Gutierrez H, Arnold RJ, Zueco J. Angiography and Optical Coherence Tomography Assessment of the Drug-Coated Balloon ESSENTIAL for the Treatment of In-Stent Restenosis. Cardiovasc Revasc Med. 2020 Apr;21(4):508-513. doi: 10.1016/j.carrev.2019.07.021. Epub 2019 Jul 23. PMID 31401071
- [Result] Her AY, Shin ES, Chung JH, Kim YH, Garg S, Lee JM, Doh JH, Nam CW, Koo BK. Plaque modification and stabilization after paclitaxel-coated balloon treatment for de novo coronary lesions. Heart Vessels. 2019 Jul;34(7):1113-1121. doi: 10.1007/s00380-019-01346-9. Epub 2019 Jan 30. PMID 30701291
- [Result] Liu Y, Zhang YJ, Deng LX, Yin ZY, Hu T, Wang Q, Li Y, Li JY, Guo WY, Mou FJ, Tao L. 12-Month clinical results of drug-coated balloons for de novo coronary lesion in vessels exceeding 3.0 mm. Int J Cardiovasc Imaging. 2019 Apr;35(4):579-586. doi: 10.1007/s10554-018-1505-z. Epub 2019 Mar 30. PMID 30929102
- [Result] Rissanen TT, Uskela S, Eranen J, Mantyla P, Olli A, Romppanen H, Siljander A, Pietila M, Minkkinen MJ, Tervo J, Karkkainen JM; DEBUT trial investigators. Drug-coated balloon for treatment of de-novo coronary artery lesions in patients with high bleeding risk (DEBUT): a single-blind, randomised, non-inferiority trial. Lancet. 2019 Jul 20;394(10194):230-239. doi: 10.1016/S0140-6736(19)31126-2. Epub 2019 Jun 13. PMID 31204115
- [Result] Sogabe K, Koide M, Fukui K, Kato Y, Kitajima H, Akabame S, Zen K, Nakamura T, Matoba S. Optical coherence tomography analysis of late lumen enlargement after paclitaxel-coated balloon angioplasty for de-novo coronary artery disease. Catheter Cardiovasc Interv. 2021 Jul 1;98(1):E35-E42. doi: 10.1002/ccd.29435. Epub 2020 Dec 28. PMID 33369836